CLINICAL TRIAL: NCT00358631
Title: An Eight-Week, Multicenter, Double-Blind, Placebo- and Escitalopram-Controlled Study Evaluating the Efficacy and Tolerability of Two Fixed Doses of SSR149415 (250 mg Bid and 100 mg Bid) in Outpatients With Major Depressive Disorder
Brief Title: An Eight-Week Study Evaluating the Efficacy and Tolerability of Two Doses of SSR149415 in Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI5878
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2009-04-13 (Estimated); Status verified 2009-04

CONDITIONS: Depressive Disorder
Keywords: depression; antidepressive agents; controlled clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — 1-(5-chloro-1-((2,4-dimethoxyphenyl)sulfonyl)-3-(2-methoxyphenyl)-2-oxo-2,3-dihydro-1H-indol-3-yl)-4-hydroxy-N,N-dimethyl-2-pyrrolidinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SSR149415

SUMMARY:
The objective is to evaluate the efficacy and safety of two doses of SSR149415 (250 mg and 100 mg twice daily) compared to placebo and escitalopram 10 mg once daily in outpatients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder, as defined by DSM-IV criteria and confirmed by the semi-structured MINI, recurrent episode.

Exclusion Criteria:

* Total score of less than 24 on the MADRS.
* HAM-D total score less than 18.
* Duration of the current depressive episode less than 1 month or greater than 2 years.
* Patients with a history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, fluoxetine within 1 month, MAOIs within 2 weeks, other antidepressants, anxiolytics, or mood-stabilizer (lithium, anticonvulsants) within 1 week except as allowed in the protocol.

The investigator will evaluate whether there are other reasons why a patient may not participate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change from baseline to Day 56 in the 17-item Hamilton Depression Rating Scale (HAM-D) total score.

SECONDARY OUTCOMES:
The main secondary endpoints are the changes from baseline to Day 56 in the HAM-D depressed mood item, Montgomery-Asberg Depression Rating Scale (MADRS) total, and Clinical Global Impression (CGI) Severity of Illness scores.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Griebel G, Beeske S, Stahl SM. The vasopressin V(1b) receptor antagonist SSR149415 in the treatment of major depressive and generalized anxiety disorders: results from 4 randomized, double-blind, placebo-controlled studies. J Clin Psychiatry. 2012 Nov;73(11):1403-11. doi: 10.4088/JCP.12m07804. Epub 2012 Oct 16. PMID 23146246